CLINICAL TRIAL: NCT01718977
Title: Cardiovascular Health/Outcomes: Improvements Created by Exercise and Education in SCI (CHOICES)
Acronym: CHOICES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: McMaster University (Other); Toronto Rehabilitation Institute (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Andrei Krassioukov, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H12-02945
Record Dates: First submitted 2012-10-24; First posted 2012-11-01 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Spinal Cord Injury
Keywords: Intervention; Body Weight Supported Treadmill Training; Arm Cycle Ergometry Training; carotid-to-femoral pulse wave velocity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Body Weight Supported Treadmill Training (Experimental): BWSTT protocol will consist of training of individuals with complete SCI on a treadmill with a body weight support system. BWSTT is assisted by three individuals who participate in training. One trainer provides support at the hip, and one trainer at each leg. The participant will be fitted with a harness while seated in their wheelchair and then wheeled up a ramp to the treadmill. Cables attached to the harness will be used to hoist the participant into a standing position. Appropriate body weight support will be set according to the suggested Hocoma locomotor training protocol, in which weight is added until the participant is in dynamic support as indicated by the dynamic gauge on the treadmill. Dynamic support is usually indicated at the weight where participants do not have knee-buckling during a static standing position; however, this may not be observed in all severe, motor-complete SCI participants.
  Interventions: Other: Body Weight Supported Treadmill Training
- Arm Cycle Ergometry Training (Active Comparator): Arm Cycle Ergometry Training ACET will be performed on an arm-cycle ergometer against individually determined levels of resistance. Upright hand cuffs will be used so that the hand will be placed with the thumb pointing downward, and the ergometer will be positioned so that the arm never exceeded the height of the shoulder.
  The end objective is for the individual to complete 30-minutes of exercise in 2, 15-minute bouts. For safety reasons, stop criteria for individual sessions will be set and participants will have a rest period of 5 minutes and afterwards asked if they want to stop exercise, or resume the session.
  Interventions: Other: Arm Cycle Ergometry Training

INTERVENTIONS:
Other: Body Weight Supported Treadmill Training — BWSTT protocol will consist of training of individuals with complete SCI on a treadmill with a body weight support system. BWSTT is assisted by three individuals who participate in training. One trainer provides support at the hip, and one trainer at each leg. The participant will be fitted with a harness while seated in their wheelchair and then wheeled up a ramp to the treadmill. Cables attached to the harness will be used to hoist the participant into a standing position. Appropriate body weight support will be set according to the suggested Hocoma locomotor training protocol, in which weight is added until the participant is in dynamic support as indicated by the dynamic gauge on the treadmill. Dynamic support is usually indicated at the weight where participants do not have knee-buckling during a static standing position; however, this may not be observed in all severe, motor-complete SCI participants.
  Other Names: BWSTT
  Arms: Body Weight Supported Treadmill Training
Other: Arm Cycle Ergometry Training — Arm Cycle Ergometry Training ACET will be performed on an arm-cycle ergometer against individually determined levels of resistance. Upright hand cuffs will be used so that the hand will be placed with the thumb pointing downward, and the ergometer will be positioned so that the arm never exceeded the height of the shoulder.
  The end objective is for the individual to complete 30-minutes of exercise in 2, 15-minute bouts. For safety reasons, stop criteria for individual sessions will be set and participants will have a rest period of 5 minutes and afterwards asked if they want to stop exercise, or resume the session.
  Other Names: ACET
  Arms: Arm Cycle Ergometry Training

SUMMARY:
This study aims to determine whether body weight-supported treadmill training (BWSTT) has beneficial effects, over and above arm-cycle ergometry training (ACET) on indicators of cardiovascular disease (CVD) risk in individuals with severe spinal cord injury (SCI).

After SCI, the primary cause of illness and death is CVD. Currently, preventative measures focus around increasing physical activity- especially through the use of ACET. However, ACET's capacity to improve cardiovascular health is questionable. Research has demonstrated that BWSTT, an alternative form of exercise, may be capable of improving cardiovascular health in individuals with SCI.

The studies primary outcome measure is carotid-to-femoral pulse wave velocity (cfPWV) which has been shown to have prognostic value for CVD above and beyond that of other risk factors. It is hypothesised that through large muscle mass involvement and postural challenge, the physical stimuli of BWSTT will reduce cfPWV and lower CVD risk in individuals with SCI.

DETAILED DESCRIPTION:
1. Purpose To determine whether body weight-supported treadmill training (BWSTT) has beneficial effects, over and above arm-cycle ergometry training (ACET), on arterial stiffness (carotid-to-femoral pulse wave velocity, cfPWV) and secondary health outcomes (cardiovascular, autonomic and metabolic indices, fitness, body composition, and quality of life) in individuals with chronic (≥ 1 year post-injury) motor-complete cervical and high-thoracic SCI.
2. Hypothesis Through large muscle mass involvement and postural challenge, the physical and metabolic stimuli of BWSTT will reduce carotid-to-femoral pulse wave velocity (cfPWV) by 1 m/s in individuals with established risk (i.e. cfPWV ≥ norm median value of age-matched able-bodied individuals).
3. Justification for the study Cardiovascular disease (CVD) is a leading cause of morbidity and mortality in the SCI population. It is most commonly attributed to decreased physical activity levels; therefore strategies for decreasing CVD risk are centred on increasing physical activity. Unfortunately, the exercise-training literature in populations with SCI is limited, making it difficult to design evidence-based exercise prescriptions. ACET is widely used by individuals with SCI, but there is limited evidence on its ability to improve cardiovascular health. Given the evidence linking cardiovascular measures, specifically cfPWV, and CVD risk, an exercise prescription, which is capable of eliciting both acute cardiovascular responses and chronic cardiovascular adaptations, is crucial. BWSTT has demonstrated favorable cardiovascular adaptations, but is primarily employed in individuals with incomplete SCI due to the nature of the exercise. While preliminary evidence in individuals with complete SCI suggest it may have favorable training effects, its effectiveness in a large sample of individuals with chronic, motor-complete, severe SCI has yet to be established.
4. Objectives Cardiovascular adaptations in individuals with SCI predispose them to complex secondary health problems. This study will use a comprehensive assessment of cardiovascular risk factors and two different exercise interventions to assist in developing cardiovascular risk profiles and determining if BWSTT has greater efficacy than traditional exercise interventions (ACET) for decreasing cardiovascular risk in individuals with high, severe SCI.
5. Research Method This study will employ a prospective, multi-centre, randomized, controlled, single-blinded clinical trial. A total of 60 participants (20 per site) between 18-60 years of age who have sustained a motor-complete (i.e., C4-T6, AIS A or B) traumatic SCI ≥ 1 year prior will be recruited. Only individuals with cfPWV ≥ norm median value of age-matched able-bodied individuals will be eligible to participate. The primary outcome measure (cfPWV), and secondary cardiovascular and autonomic parameters will be assessed using a combination of electrocardiography, ultrasound, blood pressure, and applanation tonometry techniques. Fitness will be determined using a peak oxygen consumption test on a arm-cycle ergometer. Body composition will be determined using a dual energy x-ray absorbitrometry (DXA) scan. Metabolic indices will be determined from blood sampling. Lastly, quality of life and physical activity levels will be assessed using questionnaires. Measurements will take place at baseline (via participation in Study 1), and 3 and 6-months of exercise training. Training will involve 3, 30 - 60 minute exercise sessions per week, for 24 weeks. Both BWSTT and ACET sessions will take place at the Blusson Spinal Cord Centre at International Collaboration On Repair Discoveries (ICORD).

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years of age
* Motor-complete SCI (AIS A or B)
* Severe SCI (C4-T6)
* Individuals must be competent to give informed consent.
* cfPWV above median for age:

  1. < 30 years = 6.1 m/s
  2. 30-39 years = 6.4 m/s
  3. 40-49 years = 6.9 m/s
  4. 50-59 years = 8.1 m/s
  5. ≥ 60 years = 9.7 m/s

Exclusion Criteria:

* History and/or symptoms of CVD or cardiopulmonary problems/disease.
* Major trauma or surgery within the last 6 months.
* Active Stage 3 or 4 pressure ulcer (based on the National Pressure Ulcer Advisory Panel classification)
* Recent (within 1 year) history of lower-extremity or non-union fracture
* Any unstable medical/psychiatric condition or substance abuse disorder that is likely to affect their ability to complete this study.
* Individuals with active medical issues such as pressure sores, urinary tract infections, hypertension, or heart disorders.
* Any cognitive dysfunction or language barrier that would prevent subjects from following English instructions.
* Subjects may be excluded at the discretion of the principal investigator due to other, unforeseen, safety issues.
* Weighing >135 kg (absolute weight capacity of the body weight-supported treadmill).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2019-10-17 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
The effect of Body Weight Support Treadmill Training (BWSTT) on carotid-to-femoral pulse wave velocity (cfPWV) in people with Spinal Cord Injury (SCI) at 3- and 6-months of exercise. | cfPWV assessed at baseline, 3- and 6-months.

SECONDARY OUTCOMES:
The effect of Body Weight Support Treadmill Training (BWSTT) on Cardiovascular parameters in people with Spinal Cord Injury (SCI) at 3- and 6-months of exercise. | Assessed at baseline, 3- and 6-months.
  Assessments of Blood Pressure & Heart Rate, Arterial Structure, Cardiac Structure & Function, Orthostatic Instability(Sit-Up Test) and 24-hr Blood Pressure Lability will be used to assess cardiovascular function.
  Parameters recorded from these tests include End Systolic Volume, End Diastolic Volume, Intraventricular Septum Systole (IVSs), Intraventricular Septum Diastole (IVSd), Left Ventricular Internal Diameter Systole (LVIDs), Left Ventricular Posterior Wall Systole (LVIDd), Left Ventricular Posterior Wall Diastole (LVPWd), Ejection Fraction, Cardiac Output, Fractional Shortening, Mitral Regurgitation (dP/dT), E/A, E/e' ratio, IVRT, DT, Lumen Diameter, Intima-Media Thickness, Wall/Lumen Ratio (Carotid, Brachial & Femoral), Systolic Blood Pressure, Diastolic Blood Pressure, Mean Arterial Blood Pressure and Heart Rate.
The effect of 6-months Body Weight Support Treadmill Training (BWSTT) on Autonomic function in people with Spinal Cord Injury (SCI). | Assessed at baseline and 6-months.
  Systolic and diastolic blood pressure, Mean Arterial Blood Pressure and Heart Rate will be measured. This outcome measure will also be assessed using the International Autonomic Standards Evaluation.
The effect of Body Weight Support Treadmill Training (BWSTT) on Body Composition in people with Spinal Cord Injury (SCI) following 6-months of exercise. | Assessed at baseline and 6-months.
  Body composition will be assessed using Dual Energy X-Ray Absorptiometry (DXA). DXA will be used to assess Height, Total Body Fat (Kg), Lean Mass (Kg), Body Fat Percentage and Bone Mineral Density. Weight, body mass index (BMI), Waist and Hip Circumferences will also be measured.
The effect of Body Weight Support Treadmill Training (BWSTT) on Metabolic and hematological parameters in people with Spinal Cord Injury (SCI) following 6-months of exercise. | Assessed at baseline and 6-months.
  Metabolic parameters will be assessed through blood analysis. Blood analysis will yield the following metabolic and hematological parameters: White Blood Cell Count, Erythrocytes, Packed Cell Volume, Hematocrit, Platelets, Hemoglobin, Red Cell Indices, glycated hemoglobin (HbA1C), Fasting Glucose, Triglycerides, Total Cholesterol, LDL-C, HDL-C, TC/HDL-C.
The effect of Body Weight Support Treadmill Training (BWSTT) on aerobic fitness in people with Spinal Cord Injury (SCI) following 6-months of exercise. | Assessed at baseline and 6-months.
  Aerobic fitness will be assessed via a VO2 Peak tests completed on an arm cycle ergometer. We will record Resting ECG, Blood Pressure, RPE, Oxygen Consumption and VO2Peak as well as feedback from the Positive and Negative Affect Scale (PANAS) and Visual Analogue Pain Scale.
The effect of Body Weight Support Treadmill Training (BWSTT) on quality of life in people with Spinal Cord Injury (SCI) at 3 months, 6 months and 12 months (6-month follow-up after the exercise intervention). | Assessed at baseline, 3 months, 6 months and 12 months (6 months following either intervention)
  Quality of life (QoL) will be assessed through questionnaires administered centrally by Dr. Kathleen Martin-Ginis of McMaster University in Hamilton, Ontario.
  Questionnaires used to assess QoL are; Leisure-Time Physical Activity, Questionnaire for People with SCI, MOS-36 Pain and Health Subscales, Autonomic Questionnaire, Satisfaction with Life Scale, Life Satisfaction Questionnaire, Self-Efficacy for Aerobic Exercise, Spinal Cord Independence Measure, Impact on Participation and Autonomy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andrei V Krassiokov, M.D., PhD, Principal Investigator — ICORD
Locations (3):
- Canada (3):
  - International Collaboration On Repair Discoveries, Vancouver, British Columbia
  - McMaster University, Hamilton, Ontario
  - Toronto Rehabilitation Institute, Toronto, Ontario

REFERENCES:
- [Background] Krassioukov AV, Currie KD, Hubli M, Nightingale TE, Alrashidi AA, Ramer L, Eng JJ, Ginis KAM, MacDonald MJ, Hicks A, Ditor D, Oh P, Verrier MC, Craven BC. Effects of exercise interventions on cardiovascular health in individuals with chronic, motor complete spinal cord injury: protocol for a randomised controlled trial [Cardiovascular Health/Outcomes: Improvements Created by Exercise and education in SCI (CHOICES) Study]. BMJ Open. 2019 Jan 4;9(1):e023540. doi: 10.1136/bmjopen-2018-023540. PMID 30612110
- [Derived] Dorey TW, Nightingale TE, Alrashidi AA, Thomas S, Currie KD, Hubli M, Balthazaar SJT, Krassioukov AV. Effects of exercise on autonomic cardiovascular control in individuals with chronic, motor-complete spinal cord injury: an exploratory randomised clinical trial. Spinal Cord. 2024 Oct;62(10):597-604. doi: 10.1038/s41393-024-01019-z. Epub 2024 Aug 31. PMID 39217247
- [Derived] Alrashidi AA, Nightingale TE, Currie KD, Hubli M, MacDonald MJ, Hicks AL, Oh P, Craven BC, Krassioukov AV. Exercise Improves Cardiorespiratory Fitness, but Not Arterial Health, after Spinal Cord Injury: The CHOICES Trial. J Neurotrauma. 2021 Nov 1;38(21):3020-3029. doi: 10.1089/neu.2021.0071. Epub 2021 Sep 3. PMID 34314235
- See also: Trial Protocol — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6326283/